CLINICAL TRIAL: NCT07319026
Title: Myeloid-derived Suppressor Cells: Characterization Of Their Role In Primary Myelofibrosis Pathogenesis For The Identification Of A New Therapeutic Target
Brief Title: Role of Myeloid-derived Suppressor Cells In Primary Myelofibrosis
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Rita Campanelli, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 2023-3.11/207
Record Dates: First submitted 2025-11-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-03

CONDITIONS: Primary Myelofibrosis (PMF); Healthy Subjects
Keywords: primary myelofibrosis; inflammation; myeloid derived suppressor cells
MeSH Terms: conditions — Primary Myelofibrosis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — * spleen tissue samples (embedded in OCT compound and snap-frozen in liquid nitrogen)
  * plasma samples (stored at -80°C)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with primary myelofibrosis (PMF): Patients with primary myelofibrosis, diagnosed according to the revised 2016 WHO classification, were enrolled at the Center for the Study of Myelofibrosis. Participants will undergo blood sampling only once during a routine visit.
- Healthy subjects: Healthy individuals participating to this study will be selected among regular blood donors at Fondazione IRCCS San Matteo. Blood samples will be taken during a blood donation.

SUMMARY:
The goals of this observational study are to investigate the role of myeloid-derived suppressor cells (MDSCs) in fueling chronic inflammation that is a relevant pathogenetic mechanism in patients with primary myelofibrosis (PMF), to study modifications in MDSC phenotype and function after treatment with JAK-inhibitors (JAK-i) and to test their participation in the neoangiogenic process. The main questions it aims to answer are:

* Do the frequency and function of MDSCs contribute to induce or sustain the inflammatory status that characterizes PMF?
* Does the number of circulating MDSCs in PMF patients correlate with clinical/biological parameters?
* Are MDSCs involved in the neoangiogenic processes that characterizes PMF?

DETAILED DESCRIPTION:
Primary myelofibrosis (PMF) is a Philadelphia-negative chronic myeloproliferative disorder characterized by: clonal expansion of a malignant hematopoietic stem cell CD34+, bone marrow (BM) fibrosis, splenomegaly, extra-medullary hematopoiesis and an extensive neoangiogenesis in BM and spleen. Ninety-five % of patients have an acquired mutation of JAK2, CALR or MPL genes determining an activation of the JAK-STAT pathway in the myeloid lineage. Inflammation is currently thought to play a relevant role in PMF pathogenesis, as proven by high levels of inflammatory cytokines with prognostic significance and by a state of chronic oxidative stress with elevated reactive oxygen species (ROS).

Myeloid-derived suppressor cells (MDSCs) are immature myeloid cells that accumulate in patients with malignancies, sepsis or chronic inflammation. In steady state, MDSCs migrate from the BM to different peripheral organs, where they differentiate into macrophages, dendritic cells or granulocytes. Cytokines and chemokines that are produced in tumor microenvironment recruit immature myeloid cells in peripheral blood (PB), spleen, liver and lymphoid organs, prevent their differentiation (through the activation of STAT3 signalling pathway) and induce their activation into MDSCs. This cell population is conventionally divided in two subsets: polymorphonuclear (PMN)- and monocytic (M)-MDSCs. Besides, MDSCs have the strong ability to reduce cytotoxic functions of T/NK cells and the potential to differentiate into endothelial cells and incorporate in tumor endothelium, favoring tumor neoangiogenesis. Finally, Wang et al. found high levels of circulating MDSCs in patients with myeloproliferative neoplasms that were able to inhibit T cell proliferation.

These premises suggest that MDSCs could have a role in the pathogenesis of PMF by inhibiting some functions of immune cells, nurturing chronic inflammation that characterizes the disease and/or boosting the angiogenesis process.

A condition of chronic inflammation is commonly associated with an increase of MDSCs (number and activity) that contributes in maintaining and fueling inflammation through induction of oxidative stress by means of ROS production. In PMF patients, inflammation is thought to play a relevant role in the pathogenesis of the disease, as proven by high levels of inflammatory cytokines with prognostic significance and by a state of chronic oxidative stress. Few years ago, Wang et al. reported in a very limited number of patients with PMF an increase of the frequency of circulating MDSCs; however, they were not able, likely due to the small size of samples, to find any correlation between the number of MDSCs and both the genetic background and the disease phenotype.

The rationale of this project stems from the observations that in PMF all the premises that favor a role for MDSCs in the pathogenesis of the disease exist: a) a status of chronic inflammation, b) a variable degree of dysfunction of the immune system (that, together with activation of the JAK/STAT pathway due to driver mutations, could be responsible of disease progression), and c) extensive neoangiogenic processes.

Based on these considerations, the investigators hypothesize that: 1) an increase in number and/or function of MDSCs is involved in the immunological dysfunction that has been described in PMF patients, 2) MDSCs, thank to their ability to acquire an endothelial phenotype and function, contribute to splenic and marrow neoangiogenesis, 3) MDSCs contribute to the maintenance of inflammation through their capacity to produce ROS and, in turn, oxidative stress at cellular level, 4) JAK-inhibitory therapy (currently the most effective symptomatic drug for reducing splenomegaly and abolish systemic symptoms in PMF) exerts its beneficial effect not only by down-regulating the JAK/STAT pathway in hematopoietic cells of patients, but also by inhibiting ROS production in MDSCs.

The significance of the project resides:

i) in the recognition of a new pathogenetic mechanism that, together and in addition to DNA mutation, contribute to the explanation of phenotypic diversity observed during the clinical course of PMF; ii) in the identification of a new target for personalized treatment of PMF.

The primary objective of this project is to investigate the role of MDSCs in fueling chronic inflammation (through the analysis of cytokines/chemokines together with their receptors), to evaluate their percentage in correlation with clinical/biological parameters, to study modifications after treatment with JAK-inhibitors (JAK-i), to test their participation in the neoangiogenic process.

Primary endpoints:

* to characterize, phenotypically and functionally, MDSC subsets (polymorphonuclear (PMN)- and monocytic (M)-MDSCs) in the PB and BM of PMF patients and healthy subjects. In case of splenectomy, we will evaluate the presence of PMN-MDSCs and M-MDSCs in spleen-derived mononuclear cells freshly obtained from patients (undergoing the procedure for therapeutic reasons) and controls (following splenectomy for traumatic lesions).
* to correlate the data with clinical and biological parameters as well as with the genotype of driver mutations of JAK2, MPL, and CALR genes in PMF patients.
* to assess, in plasma samples from PMF and controls, cytokines involved in the inflammatory process, in the immunosuppressive function, in the angiogenic activity and in the increased production of MDSCs.

Secondary endpoints are:

1. investigate if patient-derived MDSCs, cultured in proangiogenic conditions, are able to differentiate in endothelial cells angiogenic culture conditions (flow cytometry) and/or to modify their gene expression profile (by RealTime -quantitative PCR (RT-qPCR) before-, after- incubation);
2. test ex vivo the hypothesis that MDSCs are involved in the neoangiogenic processes that characterizes PMF, evaluating the presence of endothelial-like MDSCs in PMF tissues, performing immunofluorescence staining in spleen and BM sections and analyzing them by confocal microscopy;
3. verify whether MDSCs are effective targets of JAK-inhibitor drugs, testing in vitro the effects of JAK1/JAK2 inhibitors on MDSC activity and function by flow cytometry, RT-qPCR, ELISA tests.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years;
* diagnosis of primary myelofibrosis according to 2016 WHO criteria;
* willing to participate and understanding and signing the I.C.

Exclusion Criteria:

* concurrent or recent diagnosis of an inflammatory disease and/or neoplasia;
* any other condition that can confounds the ability to interpret data from the study;
* concurrent pregnancy. No vulnerable participants will be enrolled in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited at the Center for the Study of Myelofibrosis, Fondazione IRCCS Policlinico San Matteo, Pavia through referring physician.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of circulating MDSCs | From the first enrollment through study completion, an average of 1 year
  Freshly obtained PB mononuclear cells will be stained with a cocktail of 4 monoclonal antibodies, acquired on a flow cytometer and analyzed with the gating strategy set up in different papers to identify the two principal subsets of MDSCs (PMN-MDSCs and M-MDSCs). In these cells the investigators will evaluate pSTAT3, together with the ROS intracellular levels that will be detected using a commercially available kit. For all the experiments, 2x10e6 cells will be acquired on a flow cytometer FACS Canto II and analyzed using FACSDivaTM. The number of PMN-MDSCs and M-MDSCs will be calculated as percentage of the total number of acquired cells.
Correlations between MDSC and clinical/genetic parameters | From the first enrollment through study completion, an average of 1 year
  Demographic, clinical and laboratory data of PMF patients will be correlated with the percentage of circulating MDSCs.The appropriate multivariate analysis, with both categorical and continuous covariates, will be used to analyze the difference between groups. STATISTICA software (StatSoft) will be used for all statistical analyses and a P value <0.05 is considered statistically significant.

SECONDARY OUTCOMES:
Number of MDSCs in splenic tissue samples | From the first enrollment through study completion, an average of 1 year
  Slides obtained from spleen tissues OCT-embedded from PMF patients will be stained in immunochemistry or immunofluorescence to investigate MDSC presence and distribution.
Plasmatic levels of cytokines and chemokines | From the first enrollment through study completion, an average of 1 year
  Measurement of plasmatic cytokines and chemokines involved in the inflammatory process, in the immunosuppressive function, in the angiogenic activity and in the increased production of MDSCs will be performed in plasma samples obtained from PMF patients and controls. For the evaluation of each cytokine and chemokine, the investigators will utilize commercially available elisa kits, according to manifacturers' instructions. The plasmatic levels will be assessed as pg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
This observational study does not plan to make IPD because the Informed consent signed by the participants allows the Researcher to share data with other Researchers only in an aggregated form. In addition, the data will be collected and interpreted by the PI and co-workers only.

REFERENCES:
- [Background] Gangat N, Tefferi A. Myelofibrosis biology and contemporary management. Br J Haematol. 2020 Oct;191(2):152-170. doi: 10.1111/bjh.16576. Epub 2020 Mar 20. PMID 32196650
- [Background] Hasselbalch HC, Bjorn ME. MPNs as Inflammatory Diseases: The Evidence, Consequences, and Perspectives. Mediators Inflamm. 2015;2015:102476. doi: 10.1155/2015/102476. Epub 2015 Oct 28. PMID 26604428
- [Background] Koschmieder S, Chatain N. Role of inflammation in the biology of myeloproliferative neoplasms. Blood Rev. 2020 Jul;42:100711. doi: 10.1016/j.blre.2020.100711. Epub 2020 May 30. PMID 32505517
- [Background] Gabrilovich DI, Nagaraj S. Myeloid-derived suppressor cells as regulators of the immune system. Nat Rev Immunol. 2009 Mar;9(3):162-74. doi: 10.1038/nri2506. PMID 19197294
- [Background] Consonni FM, Porta C, Marino A, Pandolfo C, Mola S, Bleve A, Sica A. Myeloid-Derived Suppressor Cells: Ductile Targets in Disease. Front Immunol. 2019 May 3;10:949. doi: 10.3389/fimmu.2019.00949. eCollection 2019. PMID 31130949
- [Background] Murdoch C, Muthana M, Coffelt SB, Lewis CE. The role of myeloid cells in the promotion of tumour angiogenesis. Nat Rev Cancer. 2008 Aug;8(8):618-31. doi: 10.1038/nrc2444. Epub 2008 Jul 17. PMID 18633355
- [Background] Wang JC, Kundra A, Andrei M, Baptiste S, Chen C, Wong C, Sindhu H. Myeloid-derived suppressor cells in patients with myeloproliferative neoplasm. Leuk Res. 2016 Apr;43:39-43. doi: 10.1016/j.leukres.2016.02.004. Epub 2016 Feb 16. PMID 26943702
- [Result] Campanelli R, Carolei A, Catarsi P, Abba C, Boveri E, Paulli M, Gentile R, Morosini M, Albertini R, Mantovani S, Massa M, Barosi G, Rosti V. Circulating Polymorphonuclear Myeloid-Derived Suppressor Cells (PMN-MDSCs) Have a Biological Role in Patients with Primary Myelofibrosis. Cancers (Basel). 2024 Jul 16;16(14):2556. doi: 10.3390/cancers16142556. PMID 39061196